CLINICAL TRIAL: NCT07069790
Title: Effects of Chemotherapy Treatment on Metaboreflex, Mechanoreflex, and Baroreflex Function: PROTECT-08B Study
Acronym: PROTECT-08B
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-001
Record Dates: First submitted 2025-06-05; First posted 2025-07-17 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Breast Adenocarcinoma
Keywords: breast cancer; fatigue; muscle; heart
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test of neuromuscular fatigue and associated hemodynamic responses (Experimental)
  Interventions: Other: Test of neuromuscular fatigue and associated hemodynamic responses

INTERVENTIONS:
Other: Test of neuromuscular fatigue and associated hemodynamic responses — Baseline measurements of neuromuscular function and hemodynamic responses will be performed. Baroreflex sensitivity will be assessed using a neck collar applying positive and negative pressures to stimulate the carotid baroreceptors, thereby modulating baroreflex activity in a dose-dependent manner. Mechanoreflex activation will then be evaluated using the passive leg movement (PLM) technique. After the PLM, participants will perform four fatigue tasks, each followed by 2 minutes of post-exercise circulatory occlusion (PECO). Tasks involve isometric quadriceps contractions at 20% of maximal voluntary contraction (MVC) during 1 min (block 1), 2 min (blocks 2 and 3) and until failure (block4). Neuromuscular function will be assessed through MVC changes and quadriceps twitch responses. Mean arterial pressure (MAP) will be recorded continuously. Metaboreflex activity will be determined by plotting post-PECO changes in peripheral fatigue against the change in MAP during PECO phases.

SUMMARY:
Breast cancer is the most common cancer worldwide, with over 2.2 million new cases diagnosed in 2020. Treatments such as chemotherapy often lead to a reduced exercise capacity, mainly due to cardiovascular and neuromuscular dysfunctions. This decline appears to be primarily caused by increased central fatigue, while peripheral fatigue remains unchanged. This imbalance suggests a hyperactivation of type III-IV afferent nerve fibers, which are involved in the metaboreflex-a mechanism that significantly influences cardiovascular responses during exercise. Two non-invasive methods, post-exercise circulatory occlusion (PECO) and passive leg movement (PLM), will be used to assess this hyperactivity in patients. Additionally, baroreflex function-crucial for regulating blood pressure-will be evaluated using a direct method to determine its sensitivity and reactivity. By comparing patients with healthy controls under submaximal stimuli, this study aims to better understand chemotherapy-induced cardiovascular dysfunctions. Ultimately, the goal is to design personalized exercise programs to restore cardiovascular function and reduce treatment-related side effects.

DETAILED DESCRIPTION:
This is a cross-sectional, single-center study. It aims to compare women with breast cancer at the end of chemotherapy (Group 1 - patient group) with healthy women (with no history of cancer) matched for age, weight, and physical activity level (Group 2 - control group).

Both groups will undergo a single evaluation session lasting two hours and 25 minutes, during which cardiovascular responses and levels of neuromuscular fatigue will be assessed and compared. For the patient group, this evaluation will take place within the first three weeks following the end of chemotherapy treatment. The details and sequence of the assessments are provided in the section dedicated to the trial description.

ELIGIBILITY:
Inclusion Criteria:

Patient group :

* Stage I to III breast cancer
* Having completed (neo)adjuvant chemotherapy treatment less than three weeks ago

Control group :

- healthy women (no history of cancer) of similar age, weight, and physical activity level

Exclusion Criteria:

* History of cancer
* Any known chronic pathology
* Protected minor or adult
* Psychiatric, musculoskeletal or neurological problems
* Implantation of a pacemaker
* Pregnant woman
* Presenting at least one contraindication to the use of transient blood flow occlusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-10-02 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Characterize the metaboreflex in breast cancer patients at the end of chemotherapy treatment | 3 weeks after end of chemotherapy
  Significant difference in mean arterial pressure, in response to a submaximal exercise, at rest and during exercise, between the two groups (patients and controls)

SECONDARY OUTCOMES:
Characterize the baroreflex in breast cancer patients at the end of chemotherapy treatment. | 3 weeks after end of chemotherapy
  Significant difference in mean arterial pressure, in response to a given stimulation of the carotid baroreceptors, at rest and during exercise, between the two groups (patients and controls)
Characterize the mechanoreflex in breast cancer patients at the end of chemotherapy treatment. | 3 weeks after end of chemotherapy
  Significant difference in mean arterial pressure, in response to passive leg movement, between the two groups (patients and controls)
Compare heart rate reponses to submaximal exercise between the two groups | 3 weeks after end of chemotherapy
  Significant difference in heart rate between the two groups (patients and controls)
Compare stroke volume responses to submaximal exercise between the two groups | 3 weeks after end of chemotherapy
  Significant difference in stroke volume between the two groups (patients and controls)
Compare cardiac output reponses to submaximal exercise between the two groups | 3 weeks after end of chemotherapy
  Significant difference in cardiac output between the two groups (patients and controls)
Compare neuromuscular responses including maximal voluntary contraction (newtons), quadriceps twitch response (newtons) and voluntary activation (% of activation) levels induced by submaximal exercise between the two groups. | 3 weeks after end of chemotherapy
  Significant difference in peripheral fatigue and central fatigue between the two groups (patients and controls)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France